CLINICAL TRIAL: NCT06495463
Title: The Efficacy of Lonsurf® (Trifluridine/Tipiracil) Plus Chemotherapy in Metastatic Colorectal Cancer: Multi-center Prospective Study in Taiwan
Brief Title: Lonsurf® (Trifluridine/Tipiracil) Plus Chemotherapy in Metastatic Colorectal Cancer Prospective Study in Taiwan
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202200069A3
Record Dates: First submitted 2024-06-27; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: trifluridine/tipiracil; combination chemotherapy; metastatic colorectal cancer; irinotecan; oxaliplatin
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Irinotecan

STUDY DESIGN:
Intervention Model Description: trifluridine / tipiracil 35 mg/m2 PO twice daily on days 1-5 and day 6-14 off
  Chemotherapy (choose one) :
  oxaliplatin 85mg/m2 IV on day 1 every 14 days or irinotecan 100mg/m2 IV on day 1 every 14 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- trifluridine / tipiracil + Chemotherapy (Experimental): trifluridine / tipiracil 35 mg/m2 PO twice daily on days 1-5 and day 6-14 off
  combination with chemotherapy (choose one) : oxaliplatin 85mg/m2 IV on day 1 every 14 days or irinotecan 100mg/m2 IV on day 1 every 14 days.
  Interventions: Drug: Trifluridine/tipiracil

INTERVENTIONS:
Drug: Trifluridine/tipiracil — Trifluridine/tipiracil 35 mg/m2 PO twice daily on days 1-5 and day 6-14 off
  (choose one combination) : oxalipatin 85mg/m2 IV on day 1 every 14 days or irinotecan 100mg/m2 IV on day 1 every 14 days.
  Other Names: (choose one combination) : oxalipatin or irinotecan

SUMMARY:
Primary Endpoint : To evaluate the Disease control rate (DCR)

Secondary Endpoints:

To evaluate the Progression-free survival (PFS), Overall survival(OS) and Safety profile

DETAILED DESCRIPTION:
70 Per-protocol patients Plan to recruit 70 evaluable patients (With expected dropout rate of 22%, the sample size would be 90 subjects.) Simon's two-stage design (Simon, 1989) will be used. The null hypothesis that the true response rate is 0.45 will be tested against a one-sided alternative. In the first stage, 42 patients will be accrued. If there are 19 or fewer responses in these 42 patients, the study will be stopped. Otherwise, 28 additional patients will be accrued for a total of 70. The null hypothesis will be rejected if 39 or more responses are observed in 70 patients. This design yields a type I error rate of 0.05 and power of 0.8 when the true response rate is 0.6.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed adenocarcinoma of the metastatic colorectal cancer;
2. Previously treated with fluorouracil-, oxaliplatin-, and irinotecan-based chemotherapy, and anti-vascular endothelial growth factor (anti-VEGF) biological therapy;
3. The RAS wild-type patients need to receive anti-EGFR therapy;
4. Presence of at least one measurable tumor lesion which is defined as lesion that can be measured in at least one dimension (longest diameter) with a minimum size of : 10mm by CT scan, MRI and PET-CT(no less than double the slice thickness and a minimum of 10mm)(according to RECIST guideline version 1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2;
6. Investigators prescribe Lonsurf® for metastatic colorectal cancer patients who had prior treatment with Anti-VEGF and Anti-EGFR agent on routine basis. Depending on RAS status, patients with RAS mutant receive Lonsurf® as 3rd line treatment, those with RAS wild type receive Lonsurf® as 3rd/4th line treatment;
7. Patients received either oxaliplatin or irinotecan.

Exclusion Criteria:

1. Patients previously received Lonsurf® (Trifluridine／Tipiracil) or regorafenib;
2. With active central nervous system (CNS) metastasis (indicated by clinical symptoms, cerebral edema, steroid requirement, or progressive growth);
3. With clinically significant gastrointestinal hemorrhage;
4. Previous or current systemic malignancy with the exception of curatively treated non-melanoma skin cancer or cervical carcinoma in situ, unless there has been a disease-free interval of at least 5 years;
5. The patient at high risk from treatment complications including but not limited to symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia, uncontrolled diabetes, liver or renal failure and psychiatric illness or social situation that would preclude study compliance;
6. Active infection.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2022-03-19 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease control rate (DCR) | Tumor response will be judged according to RECIST v 1.1 criteria within every 8 weeks(± 2 week) in treatment period. The evaluation period is up to 24 months from the date of ICF is signed to first recorded progress or death whichever occurs first.
  The endpoints Disease Control Rate (DCR) is defined as the proportion of patients in whom the best overall response is determined as complete response (CR), partial response (PR) or stable disease (SD).

SECONDARY OUTCOMES:
Progression-free survival (PFS) | The evaluation period is up to 24 months from the date of ICF is signed to the date of first recorded progress.
  Progression-free survival (PFS) refers to the first treatment of trifluridine/tipiracil to disease progression or death.
Overall survival(OS) | The evaluation period is up to 48 months from the date of ICF is signed to the date of death.
  Overall survival (OS) is defined from the first treatment of Lonsurf® to death.
Safety profile | The evaluation period is up to 24 months from all adverse events occurring between the first drug intake and 30 days (inclusive) after the last administration of trial medication will be collected.
  All adverse events (AEs) will be summarized and listed. All adverse events occurring between the first drug intake and 30 days (inclusive) after the last administration of trial medication will be collected, and graded according to the common terminology criteria for adverse events (CTCAE) version 5.00.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chih Hsu, Principal Investigator — Chang Gung Memorial Hospital, Linkou, Taiwan
Locations (1):
- Chang-Gung Memorial Hospital, Linkou, Linkou District, Taiwan

REFERENCES:
- [Background] Mayer RJ, Van Cutsem E, Falcone A, Yoshino T, Garcia-Carbonero R, Mizunuma N, Yamazaki K, Shimada Y, Tabernero J, Komatsu Y, Sobrero A, Boucher E, Peeters M, Tran B, Lenz HJ, Zaniboni A, Hochster H, Cleary JM, Prenen H, Benedetti F, Mizuguchi H, Makris L, Ito M, Ohtsu A; RECOURSE Study Group. Randomized trial of TAS-102 for refractory metastatic colorectal cancer. N Engl J Med. 2015 May 14;372(20):1909-19. doi: 10.1056/NEJMoa1414325. PMID 25970050
- [Background] Temmink OH, Hoebe EK, van der Born K, Ackland SP, Fukushima M, Peters GJ. Mechanism of trifluorothymidine potentiation of oxaliplatin-induced cytotoxicity to colorectal cancer cells. Br J Cancer. 2007 Jan 29;96(2):231-40. doi: 10.1038/sj.bjc.6603549. PMID 17242697
- [Background] Temmink OH, Hoebe EK, Fukushima M, Peters GJ. Irinotecan-induced cytotoxicity to colon cancer cells in vitro is stimulated by pre-incubation with trifluorothymidine. Eur J Cancer. 2007 Jan;43(1):175-83. doi: 10.1016/j.ejca.2006.08.022. Epub 2006 Oct 16. PMID 17049227
- [Background] Argiles G, Andre T, Hollebecque A, Calvo A, Dahan L, Cervantes A, Leger C, Amellal N, Fougeray R, Tabernero J. Phase I dose-escalation of trifluridine/tipiracil in combination with oxaliplatin in patients with metastatic colorectal cancer. Eur J Cancer. 2019 May;112:12-19. doi: 10.1016/j.ejca.2019.01.101. Epub 2019 Mar 16. PMID 30889492
- [Background] Doi T, Yoshino T, Fuse N, Boku N, Yamazaki K, Koizumi W, Shimada K, Takinishi Y, Ohtsu A. Phase I study of TAS-102 and irinotecan combination therapy in Japanese patients with advanced colorectal cancer. Invest New Drugs. 2015 Oct;33(5):1068-77. doi: 10.1007/s10637-015-0271-1. Epub 2015 Jul 12. PMID 26163340
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- See also: Ministry of Health and Welfare, National Health Service. Cancer Registration Report — https://www.hpa.gov.tw/Pages/List.aspx?nodeid=269